CLINICAL TRIAL: NCT00116909
Title: A Phase II Study of Single-Agent OSI-7904L in Patients With Locally Advanced or Metastatic Squamous Cell Carcinoma of the Head and Neck Who Have Failed First-Line Therapy
Brief Title: A Study of OSI-7904L as Treatment in Patients With Head and Neck Cancer Who Have Failed First-Line Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OSI Pharmaceuticals (Industry)
Purpose: Treatment
Other Study IDs: OSI-904-203
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2007-03-14 (Estimated); Status verified 2007-03

CONDITIONS: Locally Recurrent or Metastatic Cancer of the Head and Neck; Must Have Failed First-Line Therapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — ((S)-2-(5-(1,2-dihydro-3-methyl-1-oxobenzo(f)-quinazoline-9-yl)methyl)amino-1-oxo-2-isoindolynyl)-glutaric acid

INTERVENTIONS:
Drug: OSI 7904L

SUMMARY:
Multi-center, Phase II study to evaluate the efficacy and safety of OSI-7904Lin head and neck cancer in patients who have failed first-line therapy

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed metastatic or locally recurrent SCCHN that is incurable with surgery or radiation therapy ECOG performance status 0-2 No more tha 1 prior chemotharapy regimen for metastatic or locally recurrent disease Adequate bone marrow, Hepatic and renal function. At least one target lesion greater than or equal to 20 mm.

Exclusion Criteria:

Symptomatic brain metasteses which are not stable, are not adequately controlled, are potenially life threatening or required radiation in the last 28 days Pregnant or lactating women. Concurrent anticancer therapy or other investigational drugs Patients with active or uncontrolled infections or other serious illnesses or medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85
Dates: Start 2004-08; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Stony Brook University Hospital, Stony Brook, New York
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - The Vanderbilt Cancer Center, Nashville, Tennessee